CLINICAL TRIAL: NCT02239393
Title: MEsenchymal Stem Cell Therapy for CAnadian MS Patients
Brief Title: Safety and Efficacy of Intravenous Autologous Mesenchymal Stem Cells for MS: a Phase 2 Proof of Concept Study
Acronym: MESCAMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20140368
Record Dates: First submitted 2014-09-10; First posted 2014-09-12 (Estimated); Last update posted 2020-03-04 (Actual); Status verified 2020-03

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Mesenchymal Stem Cells; MSC
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous Mesenchymal Stem Cells (Experimental): At week 0 a single infusion of either ex-vivo expanded autologous MSC or suspension media will be administered intravenously at a dose of 1 to 2 x 1000000 MSC/Kg body weight. At week 24, another infusion will be performed for cross-over re-treatment: at week 24 treatments will be reversed compared to week 0.
  Interventions: Biological: Mesenchymal Stem Cells
- Suspension media (Experimental): At week 0 a single infusion of either ex-vivo expanded autologous MSC or suspension media will be administered intravenously at a dose of 1 to 2 x 1000000 MSC/Kg body weight. At week 24, another infusion will be performed for cross-over re-treatment: at week 24 treatments will be reversed compared to week 0.
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — Mesenchymal Stem Cells in Plasma-Lyte A (Baxter) suspension media, containing 5% Human Albumin and 10% dimethylsulfoxide (DMSO, total volume of 5mL DMSO in final cell product) and autologous MSCs at a dose of 1 to 2 x 106 MSC/Kg participant's body weight at randomization.
  Matching placebo Plasma-Lyte A (Baxter) suspension media, containing 5% Human Albumin and 10% DMSO (total volume of 5mL DMSO in final cell product).

SUMMARY:
The mechanism of action of MSC relies on their ability to modulate pathogenic immune responses and provide neuroprotection through the release of anti-apoptotic, anti-oxidant and trophic factors as demonstrated by in-vitro and in-vivo preclinical studies.

Patients will be randomized to receive immediate vs. delayed treatment with either a dose equal to 1-2 millions/kg of body weight of autologous MSC, or equivalent volume of suspension media at baseline. At week 24 treatments will be reversed.

The primary outcome of this study is to evaluate:

* Treatment's safety within one year from MSC administration by measuring the number, time-frame and severity of adverse events and
* Treatment's activity in terms of reduction in total number of gadolinium-enhancing lesions (GEL) by magnetic resonance imaging (MRI) scans.

Secondary outcomes are to gain preliminary information on the efficacy of the experimental treatment in terms of combined MRI activity and clinical efficacy (incidence of relapses and disability progression).

DETAILED DESCRIPTION:
The mechanism of action of Mesenchymal Stem Cells (MSCs) relies on their ability to modulate pathogenic immune responses and provide neuroprotection through the release of anti-apoptotic, anti-oxidant and trophic factors as demonstrated by in vitro and in vivo preclinical studies.

Patients will be randomized to receive immediate vs. delayed treatment with either a dose equal to 1-2 millions/kg of body weight of autologous MSC, or equivalent volume of suspension media at baseline. At 6 months treatments will be reversed.

The primary outcome of this study is to evaluate

* treatment's safety within one year from MSC administration by measuring the the number, time-frame and severity of adverse event and
* treatment's activity in terms of reduction in the total number of contrast-gadolinium enhancing lesions (GEL) by magnetic resonance imaging (MRI) scans.

Secondary outcomes are to gain preliminary information on the efficacy of the experimental treatment in terms of combined MRI activity and clinical efficacy (incidence of relapses and disability progression).

ELIGIBILITY:
Inclusion Criteria:

* 1) Males and females with a diagnosis of MS

  1. Relapsing remitting MS (RRMS) not responding to at least 1 year of attempted therapy with one or more of the approved therapies (beta-interferon, glatiramer acetate, natalizumab, mitoxantrone, fingolimod, dimethyl fumarate, teriflunomide, alemtuzumab) as evidenced by at least one of the following:

     * i) ≥1 clinically documented relapse in past 12 months
     * ii) ≥2 clinically documented relapses in past 24 months
     * iii) ≥1 gadolinium-enhancing lesion (GEL) at MRI performed within the past 12 months
  2. Secondary progressive MS (SPMS) not responding to at least a year of attempted therapy with one or more of the approved therapies (beta-interferon, glatiramer acetate, natalizumab, mitoxantrone, fingolimod, dimethylfumarate, teriflunomide, alemtuzumab) as evidenced by both:

     * i) an increase of ≥1 EDSS point (if at randomization EDSS ≤ 5.0) or 0.5 EDSS point (if at randomization EDSS ≥ 5.5) in the past 12 months
     * ii) ≥1 clinically documented relapse or ≥ 1 gadolinium-enhancing lesion (GEL) at MRI within the past 12 months
  3. Primary progressive MS (PPMS) patients with all the following features:

     * i) an increase of ≥1 EDSS point (if at randomization EDSS ≤ 5.0) or 0.5 EDSS point (if at randomization EDSS ≥5.5), in the past 12 months
     * ii) ≥ 1 gadolinium-enhancing lesion (GEL) at MRI performed within the past 12 months
     * iii) positive cerebrospinal fluid (CSF) (oligoclonal banding)
* 2) Age 18 to 50 years old, inclusive at time of informed consent
* 3) Disease duration 2 to 15 years (inclusive)
* 4) EDSS 2.5 to 6.5
* 5) Able and willing to sign informed consent prior to any study-related activities

Exclusion Criteria:

* 1) RRMS not fulfilling inclusion criteria
* 2) SPMS not fulfilling inclusion criteria
* 3) PPMS not fulfilling inclusion criteria
* 4) A history of active or chronic infection including infection with HIV1-2, chronic Hepatitis B or Hepatitis C
* 5) Treatment with any immunosuppressive therapy, including natalizumab and fingolimod, within the 3 months prior to randomization
* 6) Previous treatment with cladribine or alemtuzumab
* 7) Treatment with interferon-beta, glatiramer acetate, teriflunomide or dimethyl fumarate within the 30 days prior to randomization (all teriflunomide patients will be required to have followed a wash-out with either cholestyramine or activated charcoal as indicated in the product monograph)
* 8) Treatment with corticosteroids within the 30 days prior to randomization
* 9) Relapse occurred during the 60 days prior to randomization
* 10) Previous history of a malignancy (patient reported) other than basal cell carcinoma of the skin or carcinoma in situ that has been in remission for more than one year
* 11) Severely limited life expectancy by any other co-morbid illness
* 12) History of previous diagnosis of myelodysplasia or previous hematologic disease (patient reported) or current clinically relevant abnormalities of white blood cell counts
* 13) Pregnancy or risk of pregnancy (this includes participants that are not willing to practice active contraception for the duration of the study)
* 14) eGFR < 60 mL/min/1.73m2 or known renal failure or inability to undergo MRI examination
* 15) Known allergy to gentamicin or related aminoglycosides
* 16) Inability to give written informed consent in accordance with research ethics board guidelines
* 17) Concomitant participation in another clinical trial
* 18) Inability to adhere to protocol according to the investigator's medical judgement

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2015-06; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Safety | 24 weeks from first infusion
  Incidence and severity of adverse events in MSC treatment group compared to placebo group
Efficacy | 24 weeks from first infusion
  Total number of gadolinium-enhancing lesions (GEL) on MRI scan

SECONDARY OUTCOMES:
Efficacy | 48 weeks from first infusion
  Number of gadolinium-enhancing lesions (GEL) counted over week 28, 36, 48 compared with the number of GEL counted over 4, 12, 24 weeks.
Efficacy | 24 weeks from first infusion
  Combined unique magnetic resonance imaging (MRI) activity (number of new or enlarging T2, or enhancing or re-enhancing lesions), volume of gadolinium-enhancing lesions (GEL) and volume of black holes (BH) over 4, 12, 24 weeks compared between treatment groups.
Efficacy | 48 weeks from first infusion
  Combined unique magnetic resonance imaging (MRI) activity, volume of gadolinium-enhancing lesions (GEL) and volume of black holes (BH) over week 28, 36, 48 compared with the same outcomes over 4, 12 and 24 weeks.
Efficacy | 48 weeks from first infusion
  Number of relapses in MSC treatment group vs. placebo group in the first 24 weeks and after cross-over re-treatment in the two groups.
Efficacy | 48 weeks from first infusion
  Time to sustained progression of disability and proportion of progression-free patients compared between treatment groups during the first 24 weeks and after cross-over.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S. Freedman, MSc MD FRCPC, Principal Investigator — Ottawa Hospital Research Institute
Locations (2):
- Canada (2):
  - Health Sciences Centre, Winnipeg, Manitoba
  - Ottawa Hospital - General Campus, Ottawa, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thebault S, Reaume M, Marrie RA, Marriott JJ, Furlan R, Laroni A, Booth RA, Uccelli A, Freedman MS. High or increasing serum NfL is predictive of impending multiple sclerosis relapses. Mult Scler Relat Disord. 2022 Mar;59:103535. doi: 10.1016/j.msard.2022.103535. Epub 2022 Jan 19. PMID 35078125
- [Derived] Uccelli A, Laroni A, Brundin L, Clanet M, Fernandez O, Nabavi SM, Muraro PA, Oliveri RS, Radue EW, Sellner J, Soelberg Sorensen P, Sormani MP, Wuerfel JT, Battaglia MA, Freedman MS; MESEMS study group. MEsenchymal StEm cells for Multiple Sclerosis (MESEMS): a randomized, double blind, cross-over phase I/II clinical trial with autologous mesenchymal stem cells for the therapy of multiple sclerosis. Trials. 2019 May 9;20(1):263. doi: 10.1186/s13063-019-3346-z. PMID 31072380